CLINICAL TRIAL: NCT04996563
Title: Patient Educational Video to Enhance Patient Decision Satisfaction for the Treatment of Pelvic Organ Prolapse
Brief Title: Patient Educational Video for Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Lisa Hickman, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021H0064
Record Dates: First submitted 2021-07-13; First posted 2021-08-09 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned prospectively to one of two interventions to evaluate the effect of the educational video intervention on their knowledge of prolapse and satisfaction in their healthcare decision making for management of prolapse.
Who Masked: Care Provider
Masking Description: Patients are asked not to unmask themselves at their visit to any staff or their care provider.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (Experimental): A brief educational video on POP will be sent electronically to participants randomized to the video group. Participants will view the video within one week prior to their consultation visit.
  Interventions: Other: Video
- No video (No Intervention): Participants assigned to this group will not be sent the educational video to view.

INTERVENTIONS:
Other: Video — A brief educational video, approximately 9 minutes in duration, on pelvic organ prolapse is sent electronically to patients to view prior to their initial visit in order to provide early access to information. The video was created to educate patients on the following key components of prolapse: the clinical condition, associated symptoms, common risk factors, evaluation and diagnosis, non-surgical treatment options, and surgical treatment options. Simple drawings and animations are included as visual aids to enhance the ability to conceptualize prolapse and its management options.
  Arms: Video

SUMMARY:
This is a single-blinded, randomized controlled trial investigating if a patient educational video on pelvic organ prolapse improves patient understanding of this pelvic floor disorder and satisfaction in their healthcare decision making for its management.

DETAILED DESCRIPTION:
This is a randomized controlled trial. Participants will be randomized either to watch a pre-visit educational video on pelvic organ prolapse (POP) in addition to routine physician counseling (intervention group) or routine physician counseling alone (control group). The counseling physician will be blinded. All participants will complete a pre-visit survey that includes the Prolapse and Incontinence Knowledge - POP (PIKQ-POP) and a demographics questionnaire. The PIKQ-POP has been validated to assess for patient knowledge of POP. Those randomized to the intervention group will take a brief survey after watching the video asking if they had any technical issues with the video and confirming they watched the video. At the end of all initial clinic visits, participants will complete a post-visit survey that includes the validated Satisfaction with Decision Scale for Pelvic Floor Disorders (SDS-PFD) to assess the primary outcome of change in patient decision satisfaction. The SDS is designed to assess satisfaction with a treatment decision. The SDS was modified into the SDS-PFD to be specific for women making decisions regarding surgical treatment for pelvic floor disorders. To assess the secondary outcomes of change in decision conflict and POP knowledge, the post-visit survey will also include a validated Decision Conflict Scale (DCS) and the PIKQ-POP. The DCS was developed to evaluate the effect of health care decision aids and decision-supporting interventions on decision uncertainty. The physician will also complete a counseling survey at the end of the visit to assess their perception of patient comprehension and their ease of counseling. After undergoing their chosen management option, participants will also complete a post-management survey in follow up which will include the SDS-PFD and PIKQ-POP.

ELIGIBILITY:
Inclusion Criteria:

* Initial evaluation for symptomatic POP
* Age greater than or equal to 18 years old
* Reliable access to text or e-mail

Exclusion Criteria:

* Pregnant women
* Presence of cognitive disability
* Non-English speaking patient or requiring interpreter assistance
* Women with a history of prior pelvic organ prolapse therapy, i.e. pelvic floor physical therapy, pessary, or surgical repair

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Difference in SDS-PFD score | Within 1 day of completion of the initial visit
  The difference in the score of a validated decision satisfaction questionnaire, the Satisfaction with Decision Scale for Pelvic Floor Disorders (SDS-PFD), will be compared between the two arms. A difference of 0.4 will be considered clinically meaningful. The SDS-PFD was modified from the original SDS to be specific for women making decisions regarding surgical treatment for PFD. It has 6 questions with a 5-point response scale. The score is calculated by taking the mean of the 6 answers (1-5). Higher scores correspond with higher satisfaction.

SECONDARY OUTCOMES:
Difference in DCS score | Within 1 day of completion of the initial visit
  The difference in the score of the Decision Conflict Scale (DCS) will be compared between the two arms. The DCS has been validated to assess decision conflict related to treatment selection. It has 16 questions. Each question is answered on a 5-point Likert scale of 0 to 4. The scores are summed, divided by 16, and multiplied by 25. Final scores range from 0 to 100 with higher scores indicating higher decision conflict.
Difference in PIKQ-POP score | Within 1 day of completion of the initial visit
  The difference in the Prolapse and Incontinence Knowledge - POP Questionnaire (PIKQ-POP) will be compared between the two arms. The PIKQ-POP has been validated to assess for patient knowledge of pelvic organ prolapse. It has 12 questions. Each correct question receives a score of 1. Each incorrect answer or answer of "I don't' know" receives a score of 0. The total score is the number of correct answers ranging from 0 to 12. Higher scores indicate higher POP knowledge.
Patient perception of their knowledge | Within 1 day of completion of the initial visit
  The difference in the patient's perception of their knowledge will be compared between the two arms. Patients will be asked their perception of their level of knowledge of pelvic organ prolapse.
Physician's perception of patient's understanding of prolapse | Within 1 day of completion of the initial visit
  The difference in the physician's perception of the patient's understanding of prolapse will be compared between the two arms. The physician will complete a counseling survey with a set of non-validated questions to assess their perception of if the patient viewed the video, the ease of counseling, and if the patient had a good understanding of their clinical issue.
Difference in SDS-PFD scores after management of prolapse | Within 2 weeks to 1 year after undergoing the chosen management option
  Patients will complete a final survey, the post-management survey. The difference in the patient's SDS-PFD scores will be compared between the two arms. The post-management survey will be administered in follow up to the patient after undergoing their chosen management option for the treatment of prolapse. Higher SDS-PDF scores correspond with higher satisfaction.
Difference in PIKQ-POP scores after management of prolapse | Within 2 weeks to 1 year after undergoing the chosen management option
  Patients will complete a final survey, the post-management survey. The difference in the patient's PIKQ-POP scores will be compared between the two arms. The post-management survey will be administered in follow up to the patient after undergoing their chosen management option for the treatment of prolapse. Higher PIKQ-POP scores indicate higher POP knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No